CLINICAL TRIAL: NCT06953570
Title: Impact of Frailty on the Median Effective Dose of Nalbuphine in Patient-Controlled Intravenous Analgesia for Postoperative Pain in Elderly Patients Undergoing Laparoscopic Gastrointestinal Surgery: A Prospective, Double-Blind, Cohort Study
Brief Title: Impact of Frailty on Nalbuphine Dose for Postoperative Analgesia in Elderly Patients Undergoing Laparoscopic GI Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Yongtao Sun (Other)
Responsible Party: Sponsor-Investigator, Yongtao Sun, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: Nalbuphine
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: PCIA; Frailty; Laparoscopic Gastrointestinal Surgery
Keywords: nalbuphine; ED50; PCIA; laparoscopic gastrointestinal surgery; frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- frailty group（F）（mFI≧0.27）: The initial PCA pump formulation for the first patient was set as: dexmedetomidine 2 μg/kg, nalbuphine 1 mg/kg, ondansetron 16 mg, diluted to 100 ml with normal saline. The study employed a modified Dixon up-and-down sequential method, with an initial dose of nalbuphine at 1 mg/kg. A resting Visual Analog Scale (VAS) score > 3 within 24 hours postoperatively was defined as a negative response. If a negative response occurred, the dose of nalbuphine for the next patient in the same group would be increased by 0.1 mg/kg (e.g., 1.0 → 1.1 mg/kg). Conversely, if a positive response occurred, the dose for the next patient would be decreased by 0.1 mg/kg (e.g., 1.0 → 0.9 mg/kg). The trial was terminated when eight consecutive negative-to-positive inflection points were observed.
- pre-frailty group (P)(0<mFI<0.27): The initial PCA pump formulation for the first patient was set as: dexmedetomidine 2 μg/kg, nalbuphine 1 mg/kg, ondansetron 16 mg, diluted to 100 ml with normal saline. The study employed a modified Dixon up-and-down sequential method, with an initial dose of nalbuphine at 1 mg/kg. A resting Visual Analog Scale (VAS) score > 3 within 24 hours postoperatively was defined as a negative response. If a negative response occurred, the dose of nalbuphine for the next patient in the same group would be increased by 0.1 mg/kg (e.g., 1.0 → 1.1 mg/kg). Conversely, if a positive response occurred, the dose for the next patient would be decreased by 0.1 mg/kg (e.g., 1.0 → 0.9 mg/kg). The trial was terminated when eight consecutive negative-to-positive inflection points were observed.
- non-frailty group (N)（mFI=0）: The initial PCA pump formulation for the first patient was set as: dexmedetomidine 2 μg/kg, nalbuphine 1 mg/kg, ondansetron 16 mg, diluted to 100 ml with normal saline. The study employed a modified Dixon up-and-down sequential method, with an initial dose of nalbuphine at 1 mg/kg. A resting Visual Analog Scale (VAS) score > 3 within 24 hours postoperatively was defined as a negative response. If a negative response occurred, the dose of nalbuphine for the next patient in the same group would be increased by 0.1 mg/kg (e.g., 1.0 → 1.1 mg/kg). Conversely, if a positive response occurred, the dose for the next patient would be decreased by 0.1 mg/kg (e.g., 1.0 → 0.9 mg/kg). The trial was terminated when eight consecutive negative-to-positive inflection points were observed.

SUMMARY:
This study aims to investigate the ED50 and ED95 of nalbuphine combined with dexmedetomidine in patient-controlled intravenous analgesia (PCIA) for elderly patients with different degrees of frailty, as well as their analgesic effects and complications. The results of this study can provide safe and effective dosage guidance for postoperative analgesia in frail patients, help optimize analgesic regimens, reduce the risk of complications, and improve the quality of postoperative recovery.

DETAILED DESCRIPTION:
With the increasing aging of the population in China, the proportion of elderly patients in the surgical population is continuously rising, with elderly frail patients accounting for as high as 25-50%. Previous studies have shown that postoperative pain management in elderly frail patients is associated with four major issues:

1. Enhanced pain perception.
2. Decreased pain tolerance.
3. Changes in pharmacokinetics and pharmacodynamics.
4. Iatrogenic titration patterns.

Patient-controlled intravenous analgesia (PCIA) is one of the most commonly used analgesic methods, which can shorten hospital stays, reduce the incidence of perioperative complications, and improve quality of life. However, elderly patients are more prone to hypotension, nausea, and vomiting, necessitating additional antiemetics and rescue analgesics. Nalbuphine, a dual-acting drug as a κ-receptor agonist and μ-receptor antagonist, has analgesic potency comparable to morphine and a longer duration of action (3-6 hours). However, studies have shown that due to reduced liver and kidney function, the metabolism of Nalbuphine is prolonged in elderly frail patients. Dexmedetomidine, a highly selective α2-receptor agonist with sedative, analgesic, anxiolytic, and sympatholytic properties, can reduce postoperative cardiovascular complications, enhance opioid analgesia, and lower the incidence of postoperative delirium, making it an ideal choice for multimodal analgesia. However, no studies have yet explored the dose-response relationship of dexmedetomidine combined with Nalbuphine in elderly frail patients, especially the impact of different degrees of frailty (such as mFI classification) on the median effective dose (ED50) of Nalbuphine.

This study, for the first time, employs the modified Dixon up-and-down sequential method to systematically evaluate the influence of different degrees of frailty on the ED50 of Nalbuphine-dexmedetomidine combination analgesia in elderly patients undergoing laparoscopic gastrointestinal surgery, and to analyze its analgesic effects and complication risks. The results of this study will provide evidence-based guidance for precise pain management in frail patients and promote the application of Enhanced Recovery After Surgery (ERAS) principles in the elderly frail population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who plan to undergo elective gastrointestinal surgery and are expected to stay in hospital for ≥3 days after surgery [except abdominal perineal combined with radical resection of rectal cancer (MILES)];
2. ASA grade I-Ⅳ;
3. Age ≥65 years (2);
4. 18.5 kg/m²≤BMI<30 kg/m²;
5. Sign the informed consent form.

Exclusion Criteria:

1. Severe cardiopulmonary, liver, kidney and coagulation dysfunction
2. Chemotherapy and radiotherapy were administered 1 month before surgery, and sedatives, antiemetic or antipruritic drugs were administered 24 hours before surgery
3. History of drug abuse, chronic pain, mental illness, or allergy to the drugs used in this study
4. Plan postoperative intubation or transfer to ICU;
5. Participated in other clinical studies within the past 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing laparoscopic gastrointestinal surgery
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Median Effective Dose (ED50) of Nalbuphine Based on Visual Analogue Scale (VAS) for Resting Pain at 24 Hours After Surgery | Within 24 hours after the end of surgery
  The median effective dose (ED50) of nalbuphine is defined as the dose at which 50% of patients report a resting Visual Analogue Scale (VAS) pain score of ≤3 within 24 hours postoperatively. The VAS is a 10-cm line scale ranging from 0 (no pain) to 10 (worst imaginable pain), evaluated at rest.

SECONDARY OUTCOMES:
Dose of Nalbuphine Required to Achieve Resting VAS ≤3 in 95% of Patients Within 24 Hours After Surgery (ED95) | Within 24 hours after the end of surgery
  The 95% effective dose (ED95) of nalbuphine is defined as the dose at which 95% of patients report a resting pain score of ≤3 on the Visual Analogue Scale (VAS) within 24 hours after laparoscopic gastrointestinal surgery. The VAS is a 10-cm horizontal line scale from 0 (no pain) to 10 (worst pain imaginable), evaluated in a supine resting state
Resting/Moving VAS (VASR/ VASM) | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  The VAS is assessed at rest and during moving (coughing or changing position from back to side in bed). The pain degree was assessed with a 10cm scale (0-10 points) : 0 was no pain; A score below 3 indicates mild pain, which the patient can tolerate; 4-6 patients pain and affect sleep, can still tolerate; 7-10 points patients have gradually intense pain, the pain is unbearable.
Ramsay Sedation Score (RASS) | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  1 awake, patient anxious, restless or irritable; 2 points awake, patient cooperation, good orientation or quiet; At 3 points of wakefulness, the patient only responds to commands; 4 minutes sleep, patients respond quickly to tapping eyebrow or Johnson stimulation; 5 minutes sleep, the patient is slow to tap eyebrow or Johnson stimulation; 6 minutes of sleep, the person did not respond to tapping the eyebrow or Johnson stimulation.
Brinell comfort Scale (BCS) | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  0 is persistent pain; 1 is painless at rest, severe pain when breathing deeply or coughing; 2 are painless at rest, mild pain when breathing deeply or coughing; There was no pain during 3 minutes of quiet and deep breathing. 4 points: No pain when coughing.
Nausea and vomiting (PONV) | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  Nausea is an uncomfortable feeling of wanting to vomit, but there is no contractive movement of the abdominal muscles, diaphragm muscles, etc. Vomiting refers to the contraction of the diaphragm, chest muscles and abdominal wall muscles, which may be accompanied by vomiting of stomach contents, including dry heaving. If the vomiting events are more than 1 minute apart, they are considered separate episodes. 0 degree indicates no nausea or vomiting. Grade I is nausea and no vomiting; Grade Ⅱ was nausea with mild vomiting; Degree III is severe vomiting requiring further treatment; Grade IV is vomiting that is difficult to control.
the effective pressing number of PCIA | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  The effective number of PCIA compressions performed by the patient after surgery
the cumulative pressing number of PCIA | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  The total number of postoperatively applied PCIA
sufentanil dose | Exiting PACU immediately
  rescue sufentanil doses in PACU
Time to recovery | Exiting PACU immediately
  length of stay in PACU
Postoperative Functional Recovery Milestones at Hospital Discharge | At hospital discharge, typically within 3 to 7 days after surgery
  Functional recovery is defined as the ability of the patient to (1) independently get out of bed, (2) walk at least 10 meters with or without assistance, (3) tolerate oral intake (clear fluids or diet), and (4) urinate spontaneously. Recovery is assessed using a standardized checklist by the attending physician or nurse prior to discharge.
Rescue Analgesic Requirements Within 48 Hours After Surgery | At 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  Number of additional doses of rescue analgesics administered to the patient within the first 48 hours postoperatively, recorded by nursing staff
Systolic Blood Pressure (SBP) Within 48 Hours After Surgery | At PACU discharge, and at 6, 12, 18, 24, 36, and 48 hours after surgery
  SBP will be measured using automated patient monitors at predefined time points. The values will be recorded and analyzed as a continuous variable.
Number of Participants Experiencing Respiratory Depression (RR <8/min or SpO₂ ≤90%) After Surgery | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  Respiratory depression is defined as a respiratory rate <8 breaths per minute or an oxygen saturation (SpO₂) ≤90% on room air. The incidence will be recorded at each predefined time point by nursing staff using bedside monitors
Number of Participants Requiring Antipruritic Medication for Persistent Itching After Surgery | At PACU discharge (immediately after anesthesia recovery), and at 6, 12, 18, 24, 36, and 48 hours after the end of surgery
  Pruritus is defined as persistent itching that leads to administration of antipruritic medication (e.g., antihistamines or corticosteroids). The number of participants requiring such medications at each time point will be recorded by medical staff.
Diastolic Blood Pressure (DBP) Within 48 Hours After Surgery | At PACU discharge, and at 6, 12, 18, 24, 36, and 48 hours after surgery
  DBP will be measured using automated patient monitors at predefined time points. The values will be recorded and analyzed as a continuous variable.
Mean Arterial Pressure (MAP) Within 48 Hours After Surgery | At PACU discharge, and at 6, 12, 18, 24, 36, and 48 hours after surgery
  MAP will be measured using automated patient monitors at each specified time point. MAP is calculated using the formula: (SBP + 2 × DBP) / 3.
Heart Rate (HR) Within 48 Hours After Surgery | At PACU discharge, and at 6, 12, 18, 24, 36, and 48 hours after surgery
  Heart rate will be measured using automated patient monitors. The values will be recorded in beats per minute (bpm) and analyzed continuously over time.
Peripheral Oxygen Saturation (SpO₂) Within 48 Hours After Surgery | At PACU discharge, and at 6, 12, 18, 24, 36, and 48 hours after surgery
  SpO₂ will be recorded using pulse oximetry. Oxygen saturation (%) will be continuously monitored and recorded at predefined intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Sun, Ph.D., Study Chair — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helme RD, Meliala A, Gibson SJ. Methodologic factors which contribute to variations in experimental pain threshold reported for older people. Neurosci Lett. 2004 May 6;361(1-3):144-6. doi: 10.1016/j.neulet.2003.12.014. PMID 15135914
- [Background] Schofield PA. The assessment and management of peri-operative pain in older adults. Anaesthesia. 2014 Jan;69 Suppl 1:54-60. doi: 10.1111/anae.12520. PMID 24303861
- [Background] Joshi GP. Multimodal analgesia techniques and postoperative rehabilitation. Anesthesiol Clin North Am. 2005 Mar;23(1):185-202. doi: 10.1016/j.atc.2004.11.010. PMID 15763418
- [Background] Yeh YC, Lin TF, Lin FS, Wang YP, Lin CJ, Sun WZ. Combination of opioid agonist and agonist-antagonist: patient-controlled analgesia requirement and adverse events among different-ratio morphine and nalbuphine admixtures for postoperative pain. Br J Anaesth. 2008 Oct;101(4):542-8. doi: 10.1093/bja/aen213. Epub 2008 Jul 17. PMID 18640992
- [Background] Pasternak GW. Molecular biology of opioid analgesia. J Pain Symptom Manage. 2005 May;29(5 Suppl):S2-9. doi: 10.1016/j.jpainsymman.2005.01.011. PMID 15907642